CLINICAL TRIAL: NCT00665405
Title: CT Study of Atelectasis After Delivery - Comparison Between Cesarian Section and Labor
Brief Title: Atelectasis During Delivery - Comparing Cesarian (c) -Section and Labor
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Joaquim Edson Vieira, Fisiopatologia Experimental FMUSP
Other Study IDs: CAP649-05
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-01

CONDITIONS: Delivery, Obstetric; Cesarean Section; Labor; Respiration Disorders; Atelectasis
Keywords: Delivery, obstetric; Atelectasis
MeSH Terms: conditions — Respiration Disorders; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PN: Control - Induced or natural labor under anesthesia
  Interventions: Radiation: CT scan
- PC: Case - Cesarean section under anesthesia
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — Thoracic CT scan

SUMMARY:
Pregnancy promotes respiratory system's restrictive component. This study observes the generation of atelectasis during labor.

DETAILED DESCRIPTION:
Pregnancy causes restriction of diaphragm movements as well as higher resistive component to the respiratory system. Spirometry studies have shown that the supine position increases risks of hypoxemia. There seems to be only casual observation regarding the generation of atelectasis during labor.

ELIGIBILITY:
Inclusion Criteria:

* post-anesthesia recovery

Exclusion Criteria:

* hemodynamic disorder during labor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hospital, obstetric division
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-07; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
atelectasis | 60-120 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo Medical School - FMUSP